CLINICAL TRIAL: NCT06340776
Title: The Effects of Acupressure on Pain, and Gastrointestinal Functions in Women With Hysterectomy: a Randomized Controlled Study
Brief Title: The Effects of Acupressure on Pain, and Gastrointestinal Functions in Women With Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, YELİZ YILDIRIM VARIŞOĞLU, Prof. Asist., Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 81321
Record Dates: First submitted 2024-03-10; First posted 2024-04-02 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Pain Management; Hysterectomy; Vomiting
MeSH Terms: conditions — Agnosia; Vomiting | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Acupressure groupThose who received acupressure application were called the experimental group, and patients who received routine post-operative care were called the control group. Acupressure application was applied to the experimental group at the third and twenty-fourth hours after surgery.
  Control group:The control group was evaluated for two days without any application.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure group (Experimental): Those who received acupressure application were called the experimental group, and patients who received routine post-operative care were called the control group. Acupressure application was applied to the experimental group at the third and twenty-fourth hours after surgery.
  Interventions: Other: Acupressure
- Control Group (No Intervention): The control group was evaluated for two days without any application.

INTERVENTIONS:
Other: Acupressure — For the acupressure application, planning was made to adjust the temperature, light and silence of the environment and to pay attention to privacy. 5 points that positively affect gastrointestinal functions and pain were selected (SP6, ST36, PC6, HT7 AND LI4). The duration of the session was determined to be approximately 18-20 minutes, depending on the preparation and pressure time to be applied on the 5 selected points (a total of 10 points were applied since each point will also be applied to its counterpart in the other extremity). Acupressure application was applied to each point for 1.5 minutes (1.5*10=15 minutes).
  Arms: Acupressure group

SUMMARY:
Aim This randomized controlled trial was conducted to evaluate the effect of acupressure application on gastrointestinal functions and pain after abdominal hysterectomy.

Materials and methods After undergoing hysterectomy, 39 women were randomised into acupressure (n=19), and control groups (n=20). Women in the acupressure group received acupressure on the mide meridian (ST36), the heart meridian (HT7), large intestine meridian (LI4), intersection of the spleen, liver and kidney meridians 6(SP6) and pericardium meridian (PC6) acupoints 30 min after admission to the clinic, for a period of 15 min, whereas those in the sham group received acupressure on locations 1-1.5 cm away from these points. The control group received standard treatment. The patient information form, Visual analog scale, the Rhodes Index of Nausea, Vomiting and Retching, and daily follow-up form were used for data collection.

DETAILED DESCRIPTION:
The study consists of two groups: control and experimental groups. Those who received acupressure application were called the experimental group, and patients who received routine post-operative care were called the control group. Acupressure application was applied to the experimental group at the third and twenty-fourth hours after surgery. The control group was evaluated without any application for two days. For the acupressure application, planning was made to adjust the temperature, light, and silence of the environment and to pay attention to privacy. 5 points that positively affect gastrointestinal functions and pain were selected (SP6, ST36, PC6, HT7, LI4). The duration of the session was determined to be approximately 18-20 minutes, depending on the preparation and pressure time to be applied on the 5 selected points (a total of 10 points were applied since each point will also be applied to its counterpart in the other extremity). Acupressure application was applied to each point for 1.5 minutes (1.5*10=15 minutes). The application was applied to a total of 39 women, 19 experimental and 20 control. No treatment was performed on the women in the control group other than routine post-operative care.

ELIGIBILITY:
Inclusion Criteria:

* women with Post hysterectomy operation
* Turkish women over the age of 18 years
* had no wounds or ulcerations in the areas where acupressure would be applied on the arms' legs
* had no intestinal obstruction, irritable bowel syndrome, inflammatory bowel disease, or abdominal herniation due to bowel cancer
* had defecated at least three times a week in the last trimester
* had stools of normal consistency; did not develop any serious postoperative complications

Exclusion Criteria:

* had chronicle constipation, fecal incontinence or diarrhea
* who used laxatives, suppositories oath enemas,
* who were immobilized,
* who did not agree to participate in the study,
* who did not speak Turkish.

Ages: 35 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Hysterectomy operation can be done in women.
Enrollment: 60 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
the score of nausea, vomiting and retching experiences | 18 month
  To evaluate the 24-hour nausea and vomiting status, the Rhodes Nausea, Vomiting and Retching Index was used to evaluate postoperative nausea and vomiting.In this scale, the number of nausea, vomiting, and retching of individuals and their distress are measured by Likert type assessment. This five-point Likert-type scale consists of eight items that measure the number and severity of nausea, vomiting, and retching in the last 24 hours. For each response, "never vomited" is scored as "0" or "never felt it", "7 or more" "severe" "more than 6 hours" "too much" is scored as 4. Items 1, 3, 6, and 7 must be reversed to score the Rhodes Index of Nausea, Vomiting, and Retching. The highest value that can be obtained from the scale is 32, meaning that as the score increases, the level of distress also increases. The scale has three subscales: symptom (nausea, vomiting, and retching) experience, occurrence, and distress.
gas output and stool formation of the participants | 18 month
  This is the form in which the patients' bowel sounds, flatulence time are defecation time are recorded for two days after hysterectomy.
postoperative pain | 18 month
  Pain intensity was evaluated with the Numerical Pain Intensity Scale, which is a single-criteria and subjective individual pain assessment method and aims to explain the severity of the patient's pain with numbers. The starting point of the scale, which consists of a horizontal line, is "0" or "no pain", and the ending point is "10" or "unbearable pain".
  There are numbers from 0 to 10 at equal intervals on the horizontal line, where 1-3 is defined as mild pain, 4-6 as moderate pain, and 7-10 as severe pain.

SECONDARY OUTCOMES:
Systolic Blood pressure | 18 month
  Postoperative vital signs was evaluated by daily following form
Heart rate | 18 month
  Postoperative vital signs was evaluated by daily following form
Diastolic blood pressure | 18 month
  Postoperative vital signs was evaluated by daily following form

CONTACTS AND LOCATIONS:
Overall Officials: MERVE YAVAŞ, Msc, Principal Investigator — Medipol University
Locations (1):
- Yeliz Yildirim Varişoğlu, Istanbul, Beykoz, Turkey (Türkiye)